CLINICAL TRIAL: NCT05942950
Title: Surgery or Casting in Older Adults With Intra-articular Distal Radius Fractures? A Surgeon Survey With Predictions of Treatment Outcomes in Older Adults
Brief Title: Predicting Outcomes of Distal Radius Fractures: a Surgeon Survey
Acronym: SSDART
Status: Completed | Type: Observational
Sponsor: JointResearch (Other)
Responsible Party: Sponsor
Other Study IDs: WO 23.056
Record Dates: First submitted 2023-07-04; First posted 2023-07-12 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Distal Radius Fractures; Survey; Distal Radius Fracture
Keywords: distal radius fracture; surgeon survey; surgeon; survey; predicting outcomes; preferences
MeSH Terms: conditions — Wrist Fractures

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this surgeon survey is to find out if orthopedic and trauma surgeons can predict outcomes in older adults with distal radius fractures. The main questions it aims to answer are:

* Can orthopedic and trauma surgeons effectively predict which treatment would benefit a patient the most in terms of good outcome versus poor outcome (based on Δ PRWE) following casting or surgical treatment for displaced intra-articular distal radius fractures?
* What are the perspectives of trauma surgeons and orthopedic surgeons on current literature?
* What factors direct trauma surgeons and orthopedic surgeons to surgery?

ELIGIBILITY:
Inclusion Criteria:

* Dutch orthopedic and trauma surgeons
* Residents
* Experience with at least five surgeries of distal radius fractures in the past 3 years

Exclusion Criteria:

* No experience with distal radius fractures

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Trauma surgeons (in training) and orthopedic surgeons (in training)
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2023-06-20 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
The percentage of correct predictions of the treatment outcome | From enrollment to the end of the data collection, up to 10 weeks
  Correct predictions of surgeons in total and per case.

CONTACTS AND LOCATIONS:
Locations (1):
- OLVG, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided